CLINICAL TRIAL: NCT01844622
Title: Clinical Applications of Domperidone in Patients With Refractory Gastroesophageal Reflux Disease or Delayed Gastric Solid-Phase Emptying
Brief Title: Clinical Applications of Domperidone in Patients With Delayed Gastric Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Responsible Party: Principal Investigator, Jamie S. Barkin, M.D., Professor of Medicine, U of Miami and Chief, Div of GI, Mt. Sinai Med. Ctr, Mt. Sinai Medical Center, Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-39-H-08
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Digestive System Disease
Keywords: Digestive System Diseases Disease
MeSH Terms: conditions — Digestive System Diseases | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Domperidone (Other): Domperidone will be given at 10 mg before each meal and at bedtime. At completion of the study, patients will receive standard medical therapy
  Interventions: Other: Domperidone

INTERVENTIONS:
Other: Domperidone — Domperidone dosage may be increased depending on how well the patient responds. However before increasing the dosage, patients will have follow-up EKG to evaluate any possible side effects including irregular heartbeats.
  Other Names: Motilium; Motillium

SUMMARY:
The purpose of the study is to treat patients with on-going slow stomach emptying(gastroesophageal reflux disease), who have failed to respond to standard therapy

DETAILED DESCRIPTION:
This is a study on the effectiveness of domperidone, which increases movement through the digestive system for relief of symptoms, in patients who have delayed gastric solid-phase emptying

ELIGIBILITY:
Inclusion Criteria:

* Persistent esophagitis
* Heartburn
* Nausea
* Vomiting
* Severe dyspepsia
* Severe chronic constipation

Exclusion Criteria:

* History of, or current arrhythmias including ventricular tachycardia, - Ventricular fibrillation and Torsade des Pointes.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-12; Primary Completion 2015-02-19 (Actual); Study Completion 2015-02-19 (Actual)

PRIMARY OUTCOMES:
Clinical Applications of Domperidone in Patients with Refractory Gastroesophageal Reflux Disease (GERD)or Delayed Gastric Solid-Phase Emptying | 5 years
  GERD or Delayed Gastric Emptying

CONTACTS AND LOCATIONS:
Overall Officials: Jamie S. Barkin, M.D., Principal Investigator — Mt. Sinai Medical Center
Locations (2):
- United States (2):
  - Division of Gastroenterology, Mt. Sinai Medical Center, Miami Beach, Florida
  - Mt. Sinai Medical Center, Division of Gastroenterology, Miami Beach, Florida